CLINICAL TRIAL: NCT01239784
Title: Neurodevelopmental Rehabilitation for Toddlers With Complex Heart Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000014278
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Heart Defects
Keywords: pediatrics; Heart Defects; Neurodevelopmental deficit; Neurodevelopmental Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental): A total of 20 children and their parents will be recruited for this study. Ten children will have had the Glenn procedure and 10 infants will have had the arterial switch operation.
  Interventions: Behavioral: Home-based neurodevelopmental rehabilitation programme

INTERVENTIONS:
Behavioral: Home-based neurodevelopmental rehabilitation programme — Participation in the study will require the parent and child to attend two assessment visits in addition to completing a series of parent and infant activities on a daily basis throughout the 10-week intervention period. The parent-led activities will include activities such as walking with the child, stacking blocks, rolling a ball to the child, hiding a toy under a blanket for the child to find, encouraging the child to kick a rattle while the child is lying on his/her back, or crawling or rolling in different directions.

SUMMARY:
The purpose of this project is to investigate the feasibility of using a home-based, parent-delivered model for providing neurodevelopmental rehabilitation programmes to infants who have had surgery for a complex heart defect.

DETAILED DESCRIPTION:
Neurodevelopmental deficits are a common morbidity among children who receive surgical treatment for complex congenital heart defects in infancy. Over 40% of children with complex heart defects will have neurodevelopmental deficits that persist throughout childhood even after a successful surgical procedure in infancy1. These deficits are typically related to basic motor perceptual motor or visual motor skills. Problems integrating what is seen (visual perceptions) with body movement (motor skills) makes it difficult for children to participate in peer play and limits their ability to succeed in school, thereby having a significant impact on the child's quality of life.

Traditional, therapist-delivered rehabilitation programmes to address these delays in neurodevelopment have not previously been attempted. It would be difficult to provide direct rehabilitation programmes to these patients given that their defects are rare and few patients are located within the same geographical area. Home-based, parent-delivered rehabilitation programmes have previously been shown to be effective at improving the motor skills of school-age children with complex heart defects5. Since a home-based parent delivered model would enable the participation of infants regardless of geographic location, the feasibility of using such a model for delivering neurodevelopmental rehabilitation should be investigated.

ELIGIBILITY:
Inclusion Criteria:

Families will be eligible to participate in this study if the child:

* Had the arterial switch operation (for transposition of the great arteries) or has had a Glenn procedure (for functional single ventricle).
* Is medically stable for normal infant activities.
* Is between 12 and 24 months of age in January 2010.

Exclusion Criteria:

Families will be excluded from study participation if:

* The child has a recognized syndrome or other disability affecting neurodevelopment.
* The child has had a medical procedure in the 3 months preceding the baseline study assessment.
* The cardiologist responsible for the child's care refuses to allow the child's participation.
* The child performs substantially above age-appropriate developmental milestones during the initial assessment (in which case an intervention is unlikely to have a detectable additional benefit).

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in child's neurodevelopmental status at four months using the Peabody Development Motor Scales | Baseline and four months
  The Peabody Development Motor Scale has demonstrated validity and reliability for children from birth to 5 years of age. Six subtests (reflexes, stationary, locomotion, object manipulation, grasping, visual-motor integration) yield gross, fine and total motor quotient scores.

SECONDARY OUTCOMES:
Parents opinion on the home-based neurodevelopmental rehabilitation programme | at 4 months
  During the final assessment, the researcher will interview the parent to obtain their perspective on delivering the study activities at home.
Research students experience and perception of guiding a home-based, parent-delivered rehabilitation programme | at 4 months
  Research students participating in this project will also be interviewed regarding their experiences and perceptions of guiding a home-based, parent-delivered rehabilitation programme.

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada